CLINICAL TRIAL: NCT02253212
Title: A Study to Evaluate the Safety of Transient Opening of the Blood-Brain Barrier by Low Intensity Pulsed Ultrasound With the SonoCloud Implantable Device in Patients With Recurrent Glioblastoma Before Chemotherapy Administration
Brief Title: Safety of BBB Opening With the SonoCloud
Acronym: SONOCLOUD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P120905; 2014-000393-19 (EudraCT Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Glioblastoma; Glioma; Brain Tumor
Keywords: Blood brain barrier (BBB); Disruption; Low intensity pulsed ultrasound (LIPU); Sonocloud device; Glioblastoma (GBM); Brain Cancer; Carboplatin; Therapeutic Ultrasound
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SonoCloud + carboplatin (Experimental): SonoCloud : dose escalation Carboplatin : min 6 cycles - individual dose determination according to renal function and AUC
  Interventions: Device: SonoCloud; Drug: Carboplatin

INTERVENTIONS:
Device: SonoCloud — SonoCloud : dose escalation
Drug: Carboplatin — Carboplatin : min 6 cycles - individual dose determination according to renal function and AUC

SUMMARY:
PURPOSE: The purpose of this study is to determine whether transient opening of the blood-brain barrier by pulsed ultrasound using the SonoCloud implantable ultrasound device is safely tolerated in patients with recurrent glioblastoma immediately before systemic delivery of carboplatin-based chemotherapy.

STUDY HYPOTHESIS: The blood-brain barrier can be safely opened using pulsed ultrasound prior to chemotherapy administration in patients with recurrent glioblastoma. Transient opening of the blood-brain barrier by pulsed ultrasound will increase the glioblastoma exposure to carboplatin-based chemotherapy and increase progression-free and overall survival in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
For patients with recurrent malignant gliomas, who have already been treated by a combination of surgery, radiation therapy and/or chemotherapy, few treatment options currently exist. Salvage therapies typically consist of systemic administration of chemotherapy agents, which have been shown to have limited effectiveness as median survival in this patient group is currently only 6 months.

One limitation to the efficacy of systemic chemotherapy in the treatment of brain tumors is the blood-brain barrier (BBB). To enhance the delivery of systemically administered chemotherapy agents to brain tumors, an implantable ultrasound device was developed that can be used to temporarily disrupt the BBB. Delivery of pulsed ultrasound, in combination with an ultrasound contrast agent, has been shown to temporarily disrupt the BBB for a duration of more than 6 hours and allow for a significantly increased penetration of systemically administered chemotherapy drugs in pre-clinical studies.

This study will evaluate the safety of temporary disruption of the BBB during carboplatin chemotherapy delivery in patients with recurrent glioblastoma. This study will also evaluate the maximum tolerated dose of ultrasound that can be used to disrupt the BBB.

The use of dynamic contrast-enhanced MRI will be evaluated for determining the extent and magnitude of BBB opening. Clinical efficacy (Survival) and radiological efficacy (Progression Free Survival) will also be evaluated as secondary endpoints.

ELIGIBILITY:
Inclusion criteria:

* Age greater than 18 years.
* Subjects with recurrent glioma who have failed standard therapy with surgery and/or treatment with radiation and temozolomide.
* Patient eligible for Carboplatin-based chemotherapy
* Contrast-enhanced tumor less than 35 mm in diameter
* No risk of cerebral herniation
* Able to tolerate pre/post procedure steroid treatment
* Social security affiliated (in France)
* Able and willing to give signed and informed consent
* Normal biological status
* Hemoglobin ≥ 10 g/dl
* Platelets ≥ 100000/mm3
* Neutrophils ≥ 1500/mm3
* Normal creatine clearance ≥ 60ml/mn
* ASAT < 3 N
* ALAT < 3 N
* Normal Bilirubin Level < 1.5 N
* Alkaline Phosphatase < 3 N
* INR < 1.5
* Prothrombin Level ≥ 70%

Exclusion criteria:

* Allergic to Iodine, Gadolinium, Xylocain
* Contra-indications to echographic contrast agent (microbubbles)
* Severe Renal insufficiency
* Hepatic insufficiency
* Possible toxic treatment for CNS
* Previously infected surgical field
* Uncontrolled epilepsy
* MRI contra-indications
* Hemostasis troubles thrombopenia <75.000, TP <60%, INR >1.5, anti-platelet or anticoagulant therapy on-going)
* Active phlebitis or active pulmonary embolism
* Pregnant or currently breast-feeding
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Safety of transient disruption of the blood-brain barrier using the SonoCloud system in patients with recurrent glioblastoma. | 12 months

SECONDARY OUTCOMES:
Maximum tolerated dose of ultrasound with the SonoCloud system for transient disruption of the BBB. | 12 months
Quantification of the disruption of the BBB by the SonoCloud system using dynamic T1 contrast-enhanced MRI. | 12 months
Progression-free survival in patients treated with the SonoCloud system in combination with carboplatin chemotherapy. | 12 months
Overall survival in patients treated with the SonoCloud system in combination with carboplatin chemotherapy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Idbaih, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetriere - Neurosurgery Department, Paris, France

REFERENCES:
- [Derived] Asquier N, Bouchoux G, Canney M, Martin C, Law-Ye B, Leclercq D, Chapelon JY, Lafon C, Idbaih A, Carpentier A. Blood-brain barrier disruption in humans using an implantable ultrasound device: quantification with MR images and correlation with local acoustic pressure. J Neurosurg. 2019 Feb 1;132(3):875-883. doi: 10.3171/2018.9.JNS182001. Print 2020 Mar 1. PMID 30717050
- [Derived] Goldwirt L, Canney M, Horodyckid C, Poupon J, Mourah S, Vignot A, Chapelon JY, Carpentier A. Enhanced brain distribution of carboplatin in a primate model after blood-brain barrier disruption using an implantable ultrasound device. Cancer Chemother Pharmacol. 2016 Jan;77(1):211-6. doi: 10.1007/s00280-015-2930-5. Epub 2015 Dec 8. PMID 26645405